CLINICAL TRIAL: NCT04405882
Title: Combined Technique of Corneal Remodeling to Treat Ectasia
Brief Title: Cornea Ectasia Excimer Laser Treatment
Status: Completed | Type: Observational
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Luca Buzzonetti, Head of the Ofthalmology Departement, Bambino Gesù Hospital and Research Institute
Other Study IDs: L1
Record Dates: First submitted 2020-05-18; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Corneal Ectasia
MeSH Terms: interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: topographic guided trans epithelial excimer laser — In this retrospective study 8 eyes affected by cornea ectasia of 8 patients (mean age 31.50±14.73 years) underwent simultaneous CCR and CXL. Preoperative and 6 month postoperative uncorrected distance visual acuity (UDVC) and distance corrected visual acuity (DCVA) were measured using the Efficacy and Safety index. Objective and subjective quality of vision were respectively evaluated through preoperative and 6 month postoperative corneal morphological irregularity index (CMI), National Eye Institute Visual Function NEI-VFQ25 and NEI-VFQ39 questionnaires.
  Other Names: corneal cross linking

SUMMARY:
To evaluate efficacy, safety, objective and subjective quality of vision after treatment of cornea ectasia with transepithelial topographic guided laser simultaneous Central Corneal Remodeling (CCR) and Cross-linking (CXL).

DETAILED DESCRIPTION:
Background To evaluate efficacy, safety, objective and subjective quality of vision after treatment of cornea ectasia performed with transepithelial topographic guided laser simultaneous Central Corneal Remodeling (CCR) and Cross-linking (CXL).

Methods In this retrospective study 8 eyes of 8 patients (mean age 31.50±14.73 years) affected by cornea ectasia underwent simultaneous CCR and CXL. Preoperative and 6 month postoperative uncorrected distance visual acuity (UDVC) and distance corrected visual acuity (DCVA) were measured using the Efficacy and Safety index. Objective and subjective quality of vision were evaluated preoperatively and 6 months postoperatively using corneal morphological irregularity index (CMI), National Eye Institute Visual Function NEI-VFQ25 and NEI-VFQ39 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- keratoconus with moderate severity (Amsler-Krumeich stage I-II)

Exclusion Criteria:

* concomitant ocular disease
* concomitant systemic disease
* corneal opacities

Ages: 19 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eight eyes (2 right and 6 left eyes) of 8 patients, 5 male and 3 female (mean age 31.50±14.73, range 19 to 66 years), affected by cornea ectasia were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
quality of vision | preoperatively
  uncorrected distance visual acuity (UDVC), distance corrected visual acuity (DCVA)
quality of vision | preoperatively
  Efficacy and Safety index.
quality of vision | preoperatively
  corneal morphological irregularity index (CMI)
quality of vision | 6 months postoperatively
  uncorrected distance visual acuity (UDVC), distance corrected visual acuity (DCVA)
quality of vision | 6 months postoperatively
  Efficacy and Safety index.
quality of vision | 6 months postoperatively
  corneal morphological irregularity index (CMI)

CONTACTS AND LOCATIONS:
Locations (1):
- Luca buzzonetti, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No